CLINICAL TRIAL: NCT06562972
Title: 3D Quantification Assessment of Mandibular Bone Resorption Using STL Registration-Based Superimposition Following Removable Complete Denture Occlusal Equilibration
Brief Title: 3D Assessment of Mandibular Bone Loss Via STL Superimposition After Complete Denture Occlusal Adjustment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Shady El Naggar, Associate Professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-2
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Resorption of Mandible

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal equilibration using articulating paper (Active Comparator): The articulating paper method is a widely used technique for occlusal equilibration of complete dentures. The process begins by seating the dentures properly and using thin articulating paper to mark occlusal contacts as the patient lightly bites down. High spots are identified by darker or larger marks and are carefully reduced with a fine diamond or acrylic bur. The process is repeated until even contact is achieved across all teeth. The method also involves checking occlusion during different jaw movements and making necessary adjustments. Finally, the adjusted areas are polished, and the patient's comfort is assessed.
  Interventions: Other: Occlusal equilibration of complete denture using articulating paper
- Occlusal equilibration using Occulosense (Experimental): The Oculosense system, is an advanced tool in dentistry for analyzing occlusion, especially in denture equilibration. It includes an ultra-thin sensor and software that records and displays the force and timing of occlusal contacts in real-time. This system provides detailed data on force distribution, contact timing, and the center of force, offering 2D and 3D visualizations. It allows for precise, dynamic adjustments of dentures by identifying high-pressure areas and premature contacts. Despite its benefits, including high precision and quantifiable data, it is costlier and requires specialized training.
  Interventions: Other: Occlusal equilibration of complete denture using occulosense

INTERVENTIONS:
Other: Occlusal equilibration of complete denture using articulating paper — Occlusal equilibration of complete dentures is vital for ensuring proper function, comfort, and longevity. The process aims to evenly distribute occlusal forces, eliminate premature contacts, improve stability, reduce wear, and minimize tissue trauma. It involves methods like the articulating paper technique, pressure indicator paste, T-Scan digital analysis, and clinical observation. The process includes evaluating centric and eccentric contacts, making fine adjustments, and achieving balanced articulation. Regular follow-ups are essential to monitor occlusion and make necessary adjustments, contributing to patient satisfaction and denture lifespan.
  Arms: Occlusal equilibration using articulating paper
Other: Occlusal equilibration of complete denture using occulosense — Occulosense denture equilibration is a digital occlusal analysis technique used to optimize denture fit and function. It employs a thin sensor placed between the dentures to measure bite force and timing. The system provides real-time data on occlusal contacts, allowing dentists to identify and adjust pressure points precisely. This process ensures even distribution of bite forces, enhancing denture stability, comfort, and longevity. T-Scan equilibration can significantly improve patient satisfaction by reducing pain, increasing chewing efficiency, and minimizing denture-related issues like sore spots and uneven wear.
  Arms: Occlusal equilibration using Occulosense

SUMMARY:
STL registration-based superimposition is an advanced technique for assessing mandibular bone resorption in removable complete denture (RCD) patients. This 3D method involves aligning and comparing digital models of the mandible before and after RCD use, offering high accuracy and comprehensive analysis. The process includes 3D scanning, STL conversion, registration, superimposition, and quantification. Occlusal equilibration of RCDs plays a crucial role in distributing masticatory forces and influencing bone resorption patterns. Studies using this technique have revealed non-uniform resorption, with variations in different regions of the mandible. While offering numerous advantages over traditional methods, challenges include potential registration errors and the need for specialized equipment and expertise. Future developments may incorporate machine learning, biomechanical modeling, and long-term studies to enhance understanding and clinical application of this technology in prosthodontics and oral surgery.

DETAILED DESCRIPTION:
STL registration-based superimposition is an innovative technique for evaluating mandibular bone resorption in patients using removable complete dentures (RCDs). This 3D method aligns and compares digital mandible models from different time points, providing precise volumetric and surface change measurements. The process involves 3D scanning, STL file conversion, model registration, superimposition, and quantification.

Occlusal equilibration of RCDs is crucial for distributing masticatory forces evenly, influencing bone resorption patterns. Research using this technique has shown that mandibular bone resorption is non-uniform, with variations across different mandibular regions.

While offering superior accuracy and comprehensive analysis compared to traditional methods, this approach faces challenges such as potential registration errors and the need for specialized equipment and expertise. Future developments may incorporate machine learning, biomechanical modeling, and longitudinal studies to enhance understanding and clinical application in prosthodontics and oral surgery.

ELIGIBILITY:
Inclusion Criteria

* Completely edentulous patients ranging from age 45 to 75 years
* Angle's Class I skeletal relationship
* Normal facial symmetry
* Cooperative patients
* Adequate inter-arch space not less than 12mm

Exclusion Criteria

* Temporomandibular disorders
* Uncontrolled diabetes
* Bleeding disorders or anticoagulant therapy
* Flabby tissues or sharp mandibular residual ridge.
* Heavy smokers.
* Patient's with neuromuscular disorders
* Patients on chemotherapy or radiotherapy
* Severe psychiatric disorders
* Angle's class II and III skeletal relationship

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients were excluded in the study
Enrollment: 20 (Actual)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
3D Quantification Assessment of Mandibular Bone Resorption | Baseline, thee months, six months and twelve months
  3D quantification assessment of mandibular bone resorption uses advanced imaging techniques like Cone Beam Computed Tomography (CBCT) and digital 3D software to measure and analyze bone loss in the lower jaw. This process is essential for accurate diagnosis, treatment planning (e.g., implants), and monitoring bone changes over time. It provides precise measurements, visual representations, and comprehensive analysis of bone density and volume, aiding in better clinical outcomes. Despite its advantages, it can be costly and involves radiation exposure, making it less accessible in some practices.

SECONDARY OUTCOMES:
Patient Satisfaction | Baseline, thee months, six months and twelve months
  The Oral Health Impact Profile for Edentulous Patients (OHIP-EDENT) containing 19 questions were obtained from each of the seven conceptual domains of the OHIP (functional limitation, physical pain, psychologic discomfort, physical disability, psychologic disability, social disability, and handicap)

CONTACTS AND LOCATIONS:
Overall Officials: Shady Elnaggar, Principal Investigator — Badr university in Cairo
Locations (1):
- Badr university in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No